CLINICAL TRIAL: NCT04278963
Title: Adaptive, Randomized, Single-blind, Three-arm Parallel Controlled Clinical Trial of Yinhu Qingwen Decoction in the Treatment of Mild / Common CoVID-19
Brief Title: Yinhu Qingwen Decoction for the Treatment of Mild / Common CoVID-19
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: There were no eligible patients in the paticipated centers.
Sponsor: China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Zhong Wang, Professor, China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YHQW-V3.0
Record Dates: First submitted 2020-02-19; First posted 2020-02-20 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-07

CONDITIONS: CoVID-19; Chinese Medicine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Yin Hu Qing Wen Decoction Group (Experimental): Based on the standard western medicine treatment, the patients will be given Yinhu Qingwen Decoction (Granula) for 10 days.
  Interventions: Drug: YinHu QingWen Decoction; Other: standard western medicine treatment
- Yinhu Qingwen Decoction low-dose group (Placebo Comparator): Based on the standard western medicine treatment, the patients will be given 10% dose of Yinhu Qingwen Decoction (Granula) for 10 days.
  Interventions: Drug: YinHu QingWen Decoction(low dose); Other: standard western medicine treatment
- Integrated Chinese and Western Medicine group (Active Comparator): Based on the standard western medicine treatment, the patients will be given Chinese medicine decotion granula according to their symptoms. The daily dose of Chinese medicine decoction granula will also be dissolved to 600 ml decoction and divided into 3 times(once with 200ml). The Chinese medicine decoction will be given 200ml per time, three times a day for 10 days.
  Interventions: Other: Chinese medicine treatment; Other: standard western medicine treatment

INTERVENTIONS:
Drug: YinHu QingWen Decoction — YinHu QingWen Decoction (Granula) consits of 11 Chinese herbal medicine as Honeysuckle, Polygonum cuspidatum, Schizonepeta, Longspur epimedium, etc. The decoction granula will be dissolved into 600ml decoction and divided to 3 times (once with 200ml). It will be given a 200ml per time, three times a day, for 10 days.
  Arms: Yin Hu Qing Wen Decoction Group
Drug: YinHu QingWen Decoction(low dose) — This intervention is given as 10% dose of YinHu QingWen Decoction (Granula).The granula will be dissolved into 600ml decoction and divided to 3 times (once with 200ml). It will be given a 200ml per time, three times a day, for 10 days.
  Arms: Yinhu Qingwen Decoction low-dose group
Other: Chinese medicine treatment — This intervention will be given with Chinese medicine decoction granula based on the symptoms differentiation of the patients for 10 days.
  Arms: Integrated Chinese and Western Medicine group
Other: standard western medicine treatment — Standard western medicine treatment is according to the protocol of treatment of CoVID-19 infection according to guideline appoved by National Health Commission of China.

SUMMARY:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia caused by CoVID-19, and the number of cases of infection with CoVID-19 identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally.

Given no specific antiviral therapy for CoVID-19 infection and the availability of Yinhu Qingwen Decoction as a potential antiviral Chinese medicine based on vivo antiviral studies in CoVID-19, this randomized,three-arm controlled, single-blind trial will evaluate the efficacy and safety of Yinhu Qingwen Decoction (Granula) in patients hospitalized with mild or common CoVID-19 respiratory disease.

DETAILED DESCRIPTION:
In December 2019, Wuhan, in Hubei province, China, became the center of an outbreak of pneumonia caused by CoVID-19, and the number of cases of infection with CoVID-19 identified in Wuhan increased markedly over the later part of January 2020, with cases identified in multiple other Provinces of China and internationally.

The clinical spectrum of CoVID-19 infection appears to be wide,including asymptomatic infection, mild upper respiratory disease, severe viral pneumonia with respiratory failure, and even death.However,there is no specific antiviral therapy for CoVID-19 infection, which provides a window of opportunity for testing candidate antiviral therapies. Previous experiences with SARS and MERS-CoV, highlight the need of the early intervention with Chinese medicine, and so as for CoVID-19 infection. The treatment of Chinese medicine for CoVID-19 infection suggested its benefits to improve of clinical outcomes, reduce the risk of disease progression, accelerate recovery, and reduce intensive supportive care and long-term hospitalization.

Yinhu Qingwen Decoction (Granula) consists of 11 common non-toxic traditional Chinese medicine such as Polygonum cuspidatum, Honeysuckle, Nepeta, Ligustrum lucidum. Previous vivo antiviral studies showed its activity for the inbition of CoVID-19. This clinical trial is planned to evaluate the mean clinical recovery time for patients with mild and common CoVID-19 infection as the primary outcome, and to evaluate the effect of the symptoms relief and virus clearance as well as the clinical safety.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at time of signing Informed Consent Form.
2. Laboratory (RT-PCR) confirmed infection with CoVID-19.
3. Hospitalised with Fever(≥36.7℃ -axilla or oral temperature ≥ 38.0 ℃ or ≥38.6°C tympanic or rectal) and cough;
4. No difficulty swallowing oral medications.
5. Must agree not to enroll in another study of an investigational agent prior to completion of Day 28 of study.

Exclusion Criteria:

1. Allergies, known to be allergic to research drugs or drug excipients;
2. Patient weight is less than 40 kg;
3. Respiratory distress-RR≥30 / min on room air,or SPO2≤ 93%, or PaO2/FiO2 ≤300mmHg (1mmHg = 0.133kPa)
4. Shock;
5. The clinician judges that ICU monitoring treatment is needed;
6. Patients who have participated in other clinical trials within 1 month;
7. Known patients with impaired renal function (estimated creatinine clearance <60 mL / min (male: Cr (ml / min) = (140-age) × body weight (kg) / 72 × blood creatinine concentration (mg / dl); female: Cr (ml / min) = (140-age) × weight (kg) / 85 × blood creatinine concentration (mg / dl));
8. During the screening or within 24 hours before screening, patients were found to have any of the following laboratory parameter abnormalities (based on local laboratory reference range):-ALT or AST level> 5 times the upper limit of normal range (ULN) or-ALT or AST > 3 times ULN and total bilirubin levels> 2 times ULN;
9. Being pregnant or breastfeeding, or having a positive pregnancy test at the time of pre-dose inspection, or planning to become pregnant within 3 months of study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Mean clinical recovery time (hours) | up to 28 days
  The clinical recovery time is defined as the time from initiation of study treatment (active or placebo) until normalisation of fever, respiratory rate, and oxygen saturation, and alleviation of cough, sustained for at least 72 hours.
  Normalisation and alleviation criteria:
  (1) Fever: ≤36.6°C or -axilla, ≤37.2 °C oral or ≤37.8°C rectal or tympanic;(2)Respiratory rate - ≤24/minute on room air; 3) Oxygen saturation - >94% on room air; (4) Cough - mild or absent on a patient reported scale (cough symptoms score ≤ 2 points).

SECONDARY OUTCOMES:
Time to CoVID-19 RT-PCR negative in upper respiratory tract specimen | up to 28 days
Change (reduction) in CoVID-19 viral load in upper respiratory tract specimen as assessed by area under viral load curve. | up to 28 days
Time to defervescence (in those with fever at enrolment) | up to 28 days
Time to cough reported as mild or absent (in those with cough at enrolment rated severe or moderate) | up to 28 days
Time to dyspnea reported as mild or absent (on a scale of severe, moderate, mild absent, in those with dyspnea at enrollment rated as severe or moderate) | up to 28 days
Frequency of requirement for supplemental oxygen or non-invasive ventilation | up to 28 days
Frequency of respiratory progression | up to 28 days
  Defined as: SPO2≤ 93% on room air or PaO2/FiO2≤ 300mmHg and requirement for supplemental oxygen or more advanced ventilator support.
Severe case incidence | up to 28 days
  Severe case is defined as respiratory rate ≥30/minute on room air；or Oxygen saturation - ≤94% on room air；or PaO2/FiO2≤300mmHg.
Proportion of re-hospitalization or admission to ICU | up to 28 days
All-cause mortality | up to 28 days
Frequency of serious adverse events | up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhang, Principal Investigator — Jingzhou Hospital of Traditional Chinese Medicine; Jiang-Rong Huang, M.D., Principal Investigator — Yangtze University Health Science Center; Xiao-Dong Li, M.D., Principal Investigator — Hubei Hospital of Traditional Chinese Medicine
Locations (3):
- China (3):
  - Jingzhou Hospital of Traditional Chinese Medicine, Jingzhou, Hubei
  - Wuhan Leishenshan (Thunder God Mountain) Hospital/The First Affiliated Hospital of Dalian Medical University, Wuhan, Hubei
  - Xiangyang Hospital of Traditional Chinese Medicine, Xiangyang, Hubei